CLINICAL TRIAL: NCT03933800
Title: High-flow Nasal Cannula as an Alternative Intervention for Children and Adolescents With Obstructive Sleep Apnoea
Brief Title: High Flow Nasal Cannula Therapy for Childhood OSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Kate Ching Ching Chan, Associate Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HFOSA1.0
Record Dates: First submitted 2019-04-23; First posted 2019-05-01 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Obstructive Sleep Apnea
Keywords: Therapy; High flow nasal cannula; Children; Adolescents
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High flow nasal cannula (HFNC) (Experimental): High flow nasal cannula therapy
  Interventions: Device: High flow nasal cannula
- Continuous positive airway pressure (CPAP) (Active Comparator): Continuous positive airway pressure therapy
  Interventions: Device: Continuous positive airway pressure

INTERVENTIONS:
Device: High flow nasal cannula — High flow nasal cannula therapy
  Arms: High flow nasal cannula (HFNC)
Device: Continuous positive airway pressure — Continuous positive airway pressure therapy
  Arms: Continuous positive airway pressure (CPAP)

SUMMARY:
The main objective of this study is to evaluate the efficacy of high-flow nasal cannula (HFNC) therapy in children with OSA.

Children and adolescents aged 6 to 18 years old with a diagnosis of moderate-to-severe OSA requiring CPAP therapy will be recruited.

In phase 1 study, eligible subject will be recruited for HFNC therapy titration with PSG to assess treatment efficacy. After titration, if HFNC therapy is shown to be effective, the participants will be recruited into the phase 2 intervention period to evaluate the compliance and quality of life with HFNC therapy. At baseline and follow-up visits, neurobehavioural and quality of life surveys will be completed, compliance data will be obtained.

DETAILED DESCRIPTION:
Background: Obstructive sleep apnoea (OSA) is prevalent in school-aged children and is associated with significant morbidities. Poor compliance with positive airway pressure therapy remains an issue and leads to suboptimal treatment in children with OSA. Alternative therapeutic strategy is needed to manage this group of patients more effectively.

Objective: To evaluate the efficacy of high-flow nasal cannula (HFNC) therapy in children with OSA.

Hypothesis: The investigators hypothesize that HFNC therapy is effective in reducing the severity of OSA in children.

Design: A 2-phase study - phase 1 is a single arm study to evaluate the efficacy of HFNC therapy in children with OSA, phase 2 is an intervention period to evaluate the compliance and quality of life with HFNC therapy.

Subjects: 46 children and adolescents aged 6 to 18 years old with a diagnosis of moderate-to-severe OSA requiring CPAP therapy.

Methods: In phase 1 study, eligible subject will be recruited for HFNC therapy titration with PSG to assess treatment efficacy. After titration, if HFNC therapy is shown to be effective, the participants will be recruited into the phase 2 intervention period to evaluate the compliance and quality of life with HFNC therapy. At baseline and follow-up visits, neurobehavioural and quality of life surveys will be completed, compliance data will be obtained.

Primary outcome measure: Efficacy of the HFNC therapy, as defined by the change in OAHI from baseline to that with HFNC therapy.

Expected results: Efficacy data to determine whether HFNC therapy can be an alternative therapy for children with OSA.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of moderate-to-severe OSA requiring CPAP therapy (Moderate-to-severe OSA is defined as an OAHI ≥ 5 events per hour and reported history of habitual snoring of 3 nights or more per week)

Exclusion Criteria:

* Syndromal diseases;
* Cranio-facial anomalies;
* Pathological central apnoea, chronic respiratory failure or neuromuscular disease as they would require bilevel PAP;
* Secondary obesity e.g. Prader-Willi syndrome, Cushing's syndrome;
* History of pneumothorax or pneumomediastinum;
* Prior use of PAP or HFNC therapy;
* Refusal to use non-invasive ventilation.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Efficacy of the high flow nasal cannula (HFNC) therapy: the absolute change in obstructive apnea hypopnea index (OAHI) from baseline with the use of HFNC therapy | One night - titration study will be done overnight for one night to look at the improvement of OAHI from baseline to that with HFNC therapy
  The change in obstructive apnea hypopnea index (OAHI) from baseline to that on HFNC therapy: obstructive apnoea hypopnoea index is the number of obstructive apnoea or hypopnoea events per hour of total sleep time (It is not a scale, minimum is 0 events/hour, there is no maximum score)

SECONDARY OUTCOMES:
Compliance to the therapy: percentage of subjects who are adherent to the therapy | 3 months
  Percentage of subjects who are adherent to the therapy, which is defined as >70% nightly use and average usage ≥ 4 hours per night
Quality of life measures - Modified Epworth Sleepiness Scale | 3 months
  Modified Epworth Sleepiness Scale (ESS) to assess the daytime sleepiness - ESS score is the sum of the eight item scores ranging from 0 to 24, where a higher score represents greater sleepiness.
Quality of life measures - Pediatric Quality of Life Inventory | 3 months
  Pediatric Quality of Life Inventory (PedsQL) - 23-item PedsQL Generic Core Scales will measure the core dimensions of health as delineated by the World Health Organisation, as well as role functioning. Four dimensions, physical, emotional, social and school functioning, will be measured. For physical functioning, score ranges from 1 to 8. For emotional, social and school functioning, scores range from 1 to 5. Higher scores indicate better quality of life.
Quality of life measures - OSAS-18 | 3 months
  OSAS-18 is a questionnaire with composite of OSAS-related symptoms and disease-specific quality of life. Score ranges from 18 to 126; 18 - 60 indicates small impact on health-related quality of life; 60 to 80 indicates moderate impact; >80 indicates severe impact.
Neurobehavioural surveys - Child Behaviour Checklist | 3 months
  Child Behaviour Checklist is a survey of behaviour competencies that yields standardised, age-adjusted scores on internalizing, externalizing and total behaviour difficulties

CONTACTS AND LOCATIONS:
Overall Officials: Kate C Chan, MBChB, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No